CLINICAL TRIAL: NCT05598398
Title: Evaluation of Vacuum-Assisted Closure Veraflo Therapy With Cleanse Choice Dressing on Wound Healing in Patients With Pressure Sores: A Prospective, Randomized Controlled Trial
Brief Title: NPWTi on Closure of Chronic Pressure Sores
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: 3M (Industry)
Responsible Party: Principal Investigator, Robert Galiano, Associate Professor of Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00216075
Record Dates: First submitted 2022-10-20; First posted 2022-10-28 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Pressure Sore
MeSH Terms: conditions — Pressure Ulcer | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control (Wet-to-dry dressings) (Active Comparator): Subjects randomized to the control group with receive standard of care (wet-to-dry dressings) for treatment of their pressure sore.
  Interventions: Other: Standard of Care (Wet-to-dry dressings)
- Treatment (NPWT with Instillation) (Experimental): Subjects who are randomized into the treatment arm (NPWT with Instillation) will receive the V.A.C. VeraFlo™ Cleanse Choice Dressing Systems for treatment of their pressure sore.
  Interventions: Device: V.A.C.Ulta™ Negative Pressure Wound Therapy System

INTERVENTIONS:
Device: V.A.C.Ulta™ Negative Pressure Wound Therapy System — The V.A.C.Ulta™ Negative Pressure Wound Therapy System is a 510(k) - cleared, Class II device (K100657) with the following indication for use: "the V.A.C.Ulta™ Negative Pressure Wound Therapy System is an integrated wound management system that provides Negative Pressure Wound Therapy with an instillation option.
  Arms: Treatment (NPWT with Instillation)
Other: Standard of Care (Wet-to-dry dressings) — Wet-to-dry dressings
  Arms: Control (Wet-to-dry dressings)

SUMMARY:
The primary objective of this study is to assess the effectiveness of the Negative Pressure Wound Therapy system with instillation therapy (NPWTi) on closure of chronic pressure sores. This intervention will be compared to wet-to-dry dressings, which is standard of care. In this post-market, on-label study, we hope to show that the NPWTi system more effectively closes pressure sores following debridement than traditional care.

ELIGIBILITY:
Inclusion Criteria:

1. Ischial and sacral wounds at stage 3 and 4.
2. Any pressure sore that has the potential for a good seal.

Exclusion Criteria:

1. Any pressure sore that does not have potential for a good seal.
2. Patients with fecal incontinence (due to potential for pressure sore to be near the anus).
3. Patients who by the opinion of the Principal Investigator are not candidates for surgical closure (age, BMI, comorbidities, etc.).
4. Patients who are pregnant. This is standard of care for surgery anyway, and there is uncertainty of how both the surgery and intervention would affect the fetus. We therefore stress any form of birth control, abstinence, and method to prevent pregnancy for those enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Total Length of Stay | up to 3 months
  Record the number of days spent in the hospital from initial debridement (first visit with plastic surgeon) to discharge from hospital following surgery

SECONDARY OUTCOMES:
Cost Analysis | Through study completion, approximately 5 months
  Total costs of dressings, hospital stay, direct patient care and other costs involved in inpatient care.
Number of debridements | Through study completion, approximately 5 months
  Record the total number of debridements performed at the wound site throughout the duration of the study
Successful closure of pressure sores | 2 weeks and 6 weeks post-closure surgery
  Patients will be assessed for proper closure of the wound

OTHER OUTCOMES:
Proteomic analysis | 1 year post-closure surgery
  Amount of bacteria present in frozen tissue that was collected at treatment day 1 will be determined and compared between groups using a two sample t-test.
Bioburden assessment | Through study completion, approximately 5 months
  Photos of the wound will be taken with a specialized bioburden camera, which can pick up on bacterial load of the wound. Photos will be taken before debridement, after debridement, after every dressing change, and on the day of surgery.
Wound characteristic assessments | 1 year post-closure surgery
  Wound characteristics collected by the 3D imaging as well as bioburden collected by the bioburden camera will be compared between the control and study groups. Each respective comparison will involve 2 independent sample t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Galiano, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States